CLINICAL TRIAL: NCT01826864
Title: Randomized Phase III Trial to Compare the Immunodulatory Effects of Leukine vs. Saline for Early-stage Melanoma Patients Undergoing Sentinel Lymph Node Dissection
Brief Title: Sargramostim or Hypertonic Saline Before Sentinel Lymph Node Biopsy in Treating Patients With Stage IB-II Melanoma
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: No participants enrolled
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: Genzyme, a Sanofi Company (Industry); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11-002177; NCI-2013-00645 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 5R01CA120228 (NIH)
Record Dates: First submitted 2013-04-04; First posted 2013-04-09 (Estimated); Last update posted 2020-07-27 (Actual); Status verified 2018-03

CONDITIONS: Stage IB Melanoma; Stage IIA Melanoma; Stage IIB Melanoma; Stage IIC Melanoma
MeSH Terms: conditions — Melanoma | interventions — sargramostim; Granulocyte-Macrophage Colony-Stimulating Factor; Sentinel Lymph Node Biopsy; Saline Solution, Hypertonic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (sargramostim and sentinel lymph node biopsy) (Experimental): Patients receive sargramostim SC 3-5 days prior to undergoing sentinel lymph node biopsy.
  Interventions: Biological: sargramostim; Procedure: sentinel lymph node biopsy; Other: laboratory biomarker analysis
- Arm II (hypertonic saline and sentinel lymph node biopsy) (Active Comparator): Patients receive hypertonic saline SC 3-5 days prior to undergoing sentinel lymph node biopsy.
  Interventions: Procedure: sentinel lymph node biopsy; Other: laboratory biomarker analysis; Other: hypertonic saline

INTERVENTIONS:
Biological: sargramostim — Given SC
  Other Names: GM-CSF; Leukine; Prokine
  Arms: Arm I (sargramostim and sentinel lymph node biopsy)
Procedure: sentinel lymph node biopsy — Undergo sentinel lymph node biopsy
  Other Names: sentinel node biopsy
Other: laboratory biomarker analysis — Correlative studies
Other: hypertonic saline — Given SC
  Other Names: HTS
  Arms: Arm II (hypertonic saline and sentinel lymph node biopsy)

SUMMARY:
This randomized phase III trial studies sargramostim before sentinel lymph node biopsy to see how well it works compared to hypertonic saline before sentinel lymph node biopsy in treating patients with melanoma. Biological therapies, such as sargramostim, may stimulate the immune system in different ways and stop cancer cells from growing. It is not yet known whether sargramostim is more effective than hypertonic saline in treating patients with stage IB-II melanoma undergoing sentinel lymph node biopsy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine if the alterations in morphology and phenotype to the sentinel lymph nodes are reversible.

II. To determine if the restoration of the morphology or phenotype of sentinel lymph nodes results in diminished regional tumor burden.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive sargramostim subcutaneously (SC) 3-5 days prior to undergoing sentinel lymph node biopsy.

ARM II: Patients receive hypertonic saline SC 3-5 days prior to undergoing sentinel lymph node biopsy.

After completion of study treatment, patients are followed up for 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients with stage IB or II cutaneous melanoma
* Primaries on the torso, upper and lower extremities and head and neck region
* Skin biopsy performed at least 5 days and no longer than 10 weeks from the time of initial entry into the study
* Bilirubin < 2.0 ng/dl
* Creatinine < 3.0 ng/dl
* Able to understand the consent competent to sign
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1

Exclusion Criteria:

* Prior wide excision with diameter of the excision > 3 cm
* Primary melanoma arises from the eye or mucus membranes
* Clinical evidence of regional, intransit ,or distant metastases
* Second invasive melanoma
* Prior surgical procedures that would alter the drainage patterns and would prevent us from identifying sentinel lymph nodes (SN)
* Patients with primary or secondary immunodeficiencies
* Pregnancy
* Known allergy to sargramostim (GM-CSF)
* History of cardiac disease, in particular, supraventricular tachycardia

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-08-05 (Actual); Primary Completion 2017-08-08 (Actual); Study Completion 2017-08-08 (Actual)

PRIMARY OUTCOMES:
Reversal of alterations in the SN | Up to 30 days
  A series of analysis of variance (ANOVA) models will be employed.
Proportion of subjects with positive SN in each group | Up to 30 days
  The primary analysis will be a two group continuity corrected Chi-squared test. A logistic regression analysis will also be run.

SECONDARY OUTCOMES:
Disease free survival (DFS) | Up to 30 days
  A two sample t-test will be used.
Overall survival (OS) | Up to 30 days
  A two sample t-test will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Essner, Principal Investigator — Jonsson Comprehensive Cancer Center
Locations (1):
- Jonsson Comprehensive Cancer Center, Los Angeles, California, United States